CLINICAL TRIAL: NCT03745547
Title: An Exploratory,Observational, Non-interventional, Open Label, Remote Pilot Study to Assess Adherence in Study Subjects With COPD
Brief Title: An Exploratory, Observational, Non-interventional, Open Label, Remote Pilot Study to Assess Adherence in COPD Subjects
Status: Completed | Type: Observational
Sponsor: Spire, Inc. (Industry)
Collaborators: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: SP/C/007
Record Dates: First submitted 2018-11-14; First posted 2018-11-19 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Moderate Chronic Obstructive Pulmonary Disease; Severe Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Adherence to wearing a Spire wearable health monitor — Participants will wear a Spire health monitor every day for 9 months and receive weekly emails with a short survey about the participant's condition and symptoms. If participants fail to respond to this email or Spire detects that a participant is not wearing the monitor, participants will be contacted by a nurse. While participants are wearing the monitor, Spire will make sure the sensors are collecting data but will not review the data in real time. If a participant's monitor stops sending data to Spire for more than 24 hours, the participant will be contacted. If the participant is unreachable for 10 days the participant's emergency contact will be contacted. If neither the participant nor the emergency contact is reachable over 24 days the participant will be removed from the study.

SUMMARY:
The purpose of this study is to monitor adherence to a clothing-attached breathing monitor, respiratory patterns, and activity levels in COPD patients, and correlate those respiratory patterns and activity levels with patient-reported symptoms and events. To achieve this purpose, Spire will collect data from a wearable monitor that participants attach to the participant's clothing, an associated smartphone application, and completion of weekly questions. The wearable monitor and the consumer smartphone application to be used are consumer products and currently available in the market.

This study does not include clinical intervention and no doctors will be involved in this study.

No clinical tests or office visits are included in this study. All data will be collected through an online survey tool and remotely through the wearable sensors.

DETAILED DESCRIPTION:
This is an exploratory, observational, non interventional, single-arm, open label, remote pilot study involving up to 150 self-reported COPD participants. Eligible participants will wear the Spire biophysiological health monitors for a period of 9 months while the participants report symptoms on a weekly basis via brief surveys. If and when participants incur a COPD-related exacerbation which results in a medication change after hospitalization or contact with a healthcare provider, participants will report this on the weekly surveys. When this survey is read by a study nurse, the nurse will follow up with the participant by phone to conduct a post-exacerbation phone screening. This data would provide context to inform how to correlate the biosensor-sensed physiological parameters with the exacerbation self-reported data. All study participants will be remotely distributed throughout the United States.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Self-reported diagnosis of moderate to severe COPD
* >=1 self-reported COPD-related hospitalization within the previous 12 months
* Currently using an iPhone 6 or newer and willing to install the Spire smartphone app
* Willing to wear Health Tags 80% of each 24 hour period and answer the email-based self-assessments weekly for the study duration
* Willing to provide consent to participate and abide by study protocol for study duration (9 months)
* Must be able to read and understand English
* Access to Wi-Fi at home and at work, for at least 20 hours per day (and smartphone connected to Wi-Fi throughout the study duration)

Exclusion Criteria:

* Diagnosed with another medical condition that may confound the respiratory symptoms of COPD (ex: cystic fibrosis, lung cancer, bronchiectasis, idiopathic pulmonary fibrosis, or chest wall deformities).
* Diagnosed with any neurodegenerative disorder (e,g, Parkinson's, Alzheimer's or Epilepsy)
* Pregnant at the time of study or expecting to become pregnant throughout the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult moderate Chronic Obstructive Pulmonary Disease (COPD) and severe Chronic Obstructive Pulmonary Disease (COPD) as reported by participant
Sampling Method: Non-Probability Sample
Enrollment: 184 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-11 (Actual)

PRIMARY OUTCOMES:
Spire wearable health monitor physiological data collection | weekly email surveys and phone calls over a nine month period
  To evaluate the extent to which Spire wearable health monitor can capture viable data from COPD participants

SECONDARY OUTCOMES:
Participant adherence | weekly email surveys and phone calls over a nine month period
  To evaluate the daily adherence to wearing the Spire wearable health monitor in COPD participants

CONTACTS AND LOCATIONS:
Overall Officials: Neema Moraveji, PhD, Principal Investigator — Spire, Inc.
Locations (1):
- Spire, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be available to other researchers